CLINICAL TRIAL: NCT03426046
Title: Partial Pulpotomy Treatment Of Immature Permanent Molars: A Randomized Clinical Trial
Brief Title: Treatment of Immature Permanent Teeth With Three Different Pulp Capping Materials With Partial Pulpotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Didem Sakaryali (Other)
Responsible Party: Sponsor-Investigator, Didem Sakaryali, DDS, PhD, Dr, Principal investigator, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1047
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Caries, Dental
Keywords: Biodentine; Cariously exposed pulp; MTA; Partial pulpotomy; Image J Software
MeSH Terms: conditions — Dental Caries | interventions — Pulp Capping and Pulpectomy Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Biodentine (Experimental): Partial pulpotomy treatment with Biodentine
  Interventions: Procedure: Partial Pulpotomy; Drug: Pulp Capping Agents
- Calcium Hydroxide (Active Comparator): Partial pulpotomy treatment with Calcium Hydroxide
  Interventions: Procedure: Partial Pulpotomy; Drug: Pulp Capping Agents
- Mineral Trioxide Aggregate (Experimental): Partial pulpotomy treatment with Mineral Trioxide Aggregate
  Interventions: Procedure: Partial Pulpotomy; Drug: Pulp Capping Agents

INTERVENTIONS:
Procedure: Partial Pulpotomy — Partial removal of inflamed pulp tissue in cariously exposed teeth
  Other Names: Cvek Pulpotomy, Miniature Pulpotomy
Drug: Pulp Capping Agents — Biocompatible materials
  Other Names: Pulp Capping Materials

SUMMARY:
The aim of this randomized controlled trial is to compare partial pulpotomy treatments with Biodentine®, calcium hydroxide (CH) and Mineral Trioxide Aggregate (MTA) in cariously exposed asymptomatic young permanent teeth clinically and radiographically for 1 year and evaluate root developments with Image J Software Program. The null hypothesis of this study is Biodentine® will promote healing with high success rates and induce root development more than CH and MTA.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate clinical and radiographical success of three different materials in partial pulpotomy treatment. 50 patients with 54 asymptomatic, cariously exposed young permanent mandibular molar teeth were included to the study. The teeth were randomly divided into three main groups which were; calcium hydroxide, MTA and Biodentine® and finally restorated with stainless steel crowns. Pain, percussion sensitivity, palpation sensitivity of soft tissue around the tooth, root development, presence of lesion, integrity of lamina dura were evaluated clinically and radiographically during 12 months and recorded for each. Also, Image J Program with Turbo-Reg plug in was used for standardization of the radiographs and to determine the increase in root length.

ELIGIBILITY:
Inclusion Criteria:

* Deep dentine caries with pulp exposure

Exclusion Criteria:

* Pulp exposure without hemorrhage control

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Root development | 12 months
  Root length measurement in pixels with Image J Software Program

SECONDARY OUTCOMES:
Clinical Evaluation | 12 months
  Percussion sensitivity evaluation with blunt end of a dental instrument comparing with contralateral or next healthy tooth
Radiographical Evaluation | 12 months
  Integrity of lamina dura with visual evaluation of radiopaque line around the root using image plate system

CONTACTS AND LOCATIONS:
Overall Officials: Alev Alacam, DDS, PhD, Study Chair — Gazi University, Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Gazi University, Faculty of Dentistry, Department of Pediatric Dentistry, Ankara, Turkey (Türkiye)